CLINICAL TRIAL: NCT02130388
Title: The Impact of Zinc Supplementation on Innate Immunity and Patient Safety in Sepsis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow Recruitment and funds no longer available.
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Beth Y Besecker, MD, Assistant Professor of Internal Medicine, Ohio State University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2013H0127
Record Dates: First submitted 2014-04-29; First posted 2014-05-05 (Estimated); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis | interventions — Zinc

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Renal Insufficiency (Other): Based on creatinine clearance
  Interventions: Dietary Supplement: Zinc
- Renal Sufficiency (Other): Based on creatinine clearance
  Interventions: Dietary Supplement: Zinc

INTERVENTIONS:
Dietary Supplement: Zinc

SUMMARY:
Sepsis is the body's response to a life-threatening infection. This study will determine if zinc supplementation is safe to use in patients with severe sepsis or septic shock. This study will also gather preliminary information to evaluate the impact that zinc has on the immune system (the body's defense system against infection) and whether zinc can help monocytes and macrophages (specific types of cells that remove infections from the body) work more effectively.

DETAILED DESCRIPTION:
Previous research has shown that zinc supplementation reduces the length and severity of some types of medical infections (examples include the cold virus and diarrhea). Because zinc has been shown to improve the immune system's function, some doctors provide mineral supplements such as zinc to their patients in the Intensive Care Unit. However, there are no studies to show how effective zinc is or that have evaluated what dose(s) of zinc are safe in patients with severe sepsis/septic shock. Nor have studies examined if tolerable doses for septic patients can improve how the immune system functions.

If zinc is shown to improve how the immune system functions during sepsis, it could be used in the future as part of the treatment regimen for patients with sepsis.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to an Ohio State University Medical Center medical Intensive Care Unit
* ≥ 18 years
* Have consensus criteria for severe sepsis (two of four systemic inflammatory response syndrome [SIRS] signs [tachycardia, tachypnea, fever or hypothermia, leukocytosis or leukopenia]) and a known or suspected infection resulting in an organ failure (i.e. respiratory failure, renal failure, etc.)
* Patient must consent to enrollment within 36 hours of a new episode of sepsis and be able to receive supplementation within 12 hours of enrollment but not to exceed 36 hours since sepsis onset to be eligible.

Exclusion Criteria:

* Consent not available or declined,
* Prisoner, Women who are pregnant or lactating
* Chemotherapy within past 4 weeks or Absolute Neutrophil Count<500
* AIDS defining illness or Cluster of Differentiation 4 < 200
* Acute Pancreatitis or amylase/lipase > 2x normal
* Small Bowel Obstruction or GI condition preventing enteral route of feeding
* C.difficile colitis or active diarrhea
* Active vomiting or current use of Total Parenteral Nutrition within past 30 days
* Predicted ICU length of stay < 72 hours or moribund
* End Stage Renal Disease on chronic intermittent dialysis
* Previously enrolled in this zinc supplementation study or currently enrolled in another nutritional supplementation trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-05; Primary Completion 2017-10 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Toxicity will be monitored clinically for symptoms such as new vomiting or diarrhea and by serum zinc and copper levels. | 10 days
  This study consists of receiving a dose of zinc once daily while in the ICU for up to 7 days, up to four timed blood draws over the first 10 days of your hospitalization (if you remain in the hospital that long), and collecting some immune cells from your blood +/- lungs. We will review your medical chart at the time of the blood draws and again when you are getting ready for discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Beth Besecker, MD, Principal Investigator — Ohio State University
Locations (1):
- OSU Medical Center, Columbus, Ohio, United States